CLINICAL TRIAL: NCT04143425
Title: Prospective Observational Study of Imaging-based Response Prediction for Anti-angiogenic Treatment in Recurrent Glioblastomas
Brief Title: Response Prediction for Anti-angiogenic Treatment in Recurrent Glioblastoma
Status: Completed | Type: Observational
Sponsor: Ho Sung Kim (Other)
Responsible Party: Sponsor-Investigator, Ho Sung Kim, Professor, Asan Medical Center
Organization: Asan Medical Center (Other)
Other Study IDs: AsanMCHSKim_05
Record Dates: First submitted 2019-10-27; First posted 2019-10-29 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Adult Glioblastoma; Magnetic Resonance Imaging; Bevacizimab
Keywords: Recurrent Glioblastoma; Bevacizumab; Imaging
MeSH Terms: conditions — Glioblastoma | interventions — Perfusion Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Received bevacizumab treatment: Recurrent glioblastoma patients with received anti-angiogenic treatment
  Interventions: Diagnostic Test: 3-Tesla conventional magnetic resonance imaging; Diagnostic Test: Advanced imaging without contrast use; Diagnostic Test: Dynamic susceptibility contrast-weighted imaging

INTERVENTIONS:
Diagnostic Test: 3-Tesla conventional magnetic resonance imaging — T1-weighted, T2-weighted, fluid-attenuated inversion recovery, and contrast-enhanced T1-weighted imaging
Diagnostic Test: Advanced imaging without contrast use — Diffusion-weighted imaging, amide proton transfer-weighted imaging, electrical properties tomography, and 2hG-magnetic resonance spectroscopy
Diagnostic Test: Dynamic susceptibility contrast-weighted imaging — Cerebral blood volume and vessel architectural imaging parameters

SUMMARY:
This study aims to evaluate whether pre-treatment MRI can be used to predict treatment response for anti-angiogenic treatment in glioblastomas.

DETAILED DESCRIPTION:
Although overall the effects on prolonging survival in bevacizumab-treated patients is modest at best, it is still unclear whether there is not a more substantial positive effect in a subset of patients, potentially identifiable by imaging markers. Allowing for prediction of good or bad responder from anti-angiogenic therapy prior to treatment completion is important to select patients most likely to benefit from anti-angiogenic treatment.

This is a prospective observational study and no active comparator will be used. Study participants include adult patients with recurrent glioblastoma.

We hypothesized that quantifying changes in multi-modal advanced MR imaging techniques would allow early treatment response and long-term prediction in glioblastomas.

ELIGIBILITY:
Inclusion Criteria:

1. Patients had histologically confirmed glioblastoma with progression diagnosed on the basis of clinical data and MRI after standard treatment of operation, concurrent chemoradiotherapy, and adjuvant temozolomide;
2. Patients were more than 3 months from chemoradiotherapy to avoid the confounding factor of radiation necrosis (pseudoprogression);
3. Ability to understand and the willingness to sign a written informed consent document; all patients, or their legal guardians, must sign a written informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization in accordance with institutional guidelines

Exclusion Criteria:

1. Patients were not subject to therapies other than anti-angiogenic treatment, including re-operation, re-irradiation, or immunotherapies, because of the patient's clinical status and indication
2. Patients who have any type of bioimplant activated by mechanical, electronic, or magnetic means (e.g., cochlear implants, pacemakers, neurostimulators, biostimulators, electronic infusion pumps, etc), because such devices may be displaced or malfunction

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of tertiary medical center
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2020-02-06 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Progression free survival | Average 9 months
  Time from anti-angiogenic treatment until death or the first imaging report indicating worsening/progression.

SECONDARY OUTCOMES:
6-month progression | 6 month
  Pathologic confirmation following second look surgery or clinico-radiological assessment at 6-month
Overall survival | Average 12 months
  Time from anti-angiogenic treatment to death

CONTACTS AND LOCATIONS:
Overall Officials: Ho Sung Kim, M.D.,Ph.D., Principal Investigator — Department of Radiology, Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Data sharing if raw imaging data outside Korea is prohibited by Korean government. For anonymized imaging data, part of cases may be feasible on the approval of the principle investigator.

REFERENCES:
- [Background] Pope WB, Xia Q, Paton VE, Das A, Hambleton J, Kim HJ, Huo J, Brown MS, Goldin J, Cloughesy T. Patterns of progression in patients with recurrent glioblastoma treated with bevacizumab. Neurology. 2011 Feb 1;76(5):432-7. doi: 10.1212/WNL.0b013e31820a0a8a. PMID 21282590
- [Result] Ellingson BM, Gerstner ER, Smits M, Huang RY, Colen R, Abrey LE, Aftab DT, Schwab GM, Hessel C, Harris RJ, Chakhoyan A, Gahrmann R, Pope WB, Leu K, Raymond C, Woodworth DC, de Groot J, Wen PY, Batchelor TT, van den Bent MJ, Cloughesy TF. Diffusion MRI Phenotypes Predict Overall Survival Benefit from Anti-VEGF Monotherapy in Recurrent Glioblastoma: Converging Evidence from Phase II Trials. Clin Cancer Res. 2017 Oct 1;23(19):5745-5756. doi: 10.1158/1078-0432.CCR-16-2844. Epub 2017 Jun 27. PMID 28655794
- [Result] Schmainda KM, Zhang Z, Prah M, Snyder BS, Gilbert MR, Sorensen AG, Barboriak DP, Boxerman JL. Dynamic susceptibility contrast MRI measures of relative cerebral blood volume as a prognostic marker for overall survival in recurrent glioblastoma: results from the ACRIN 6677/RTOG 0625 multicenter trial. Neuro Oncol. 2015 Aug;17(8):1148-56. doi: 10.1093/neuonc/nou364. Epub 2015 Feb 2. PMID 25646027
- [Result] Park JE, Kim HS, Park KJ, Kim SJ, Kim JH, Smith SA. Pre- and Posttreatment Glioma: Comparison of Amide Proton Transfer Imaging with MR Spectroscopy for Biomarkers of Tumor Proliferation. Radiology. 2016 Feb;278(2):514-23. doi: 10.1148/radiol.2015142979. Epub 2015 Aug 19. PMID 26491847
- [Result] Emblem KE, Mouridsen K, Bjornerud A, Farrar CT, Jennings D, Borra RJ, Wen PY, Ivy P, Batchelor TT, Rosen BR, Jain RK, Sorensen AG. Vessel architectural imaging identifies cancer patient responders to anti-angiogenic therapy. Nat Med. 2013 Sep;19(9):1178-83. doi: 10.1038/nm.3289. Epub 2013 Aug 18. PMID 23955713
- [Derived] Kim M, Park JE, Yoon SK, Kim N, Kim YH, Kim JH, Kim HS. Vessel size and perfusion-derived vascular habitat refines prediction of treatment failure to bevacizumab in recurrent glioblastomas: validation in a prospective cohort. Eur Radiol. 2023 Jun;33(6):4475-4485. doi: 10.1007/s00330-022-09164-w. Epub 2022 Oct 15. PMID 36242633
- See also: Actual publication results — https://link-springer-com-ssl.libproxy.amc.seoul.kr/article/10.1007/s00330-022-09164-w
- Available data/document: Clinical Study Report — https://link-springer-com-ssl.libproxy.amc.seoul.kr/article/10.1007/s00330-022-09164-w — Vessel size and perfusion-derived vascular habitat refines prediction of treatment failure to bevacizumab in recurrent glioblastomas: validation in a prospective cohort